CLINICAL TRIAL: NCT03031717
Title: Follow-up and Survival of Cirrhotic and Non Cirrhotic Patients With Portal Vein Thrombosis Treated With Transjugular Intrahepatic Portosystemic Shunt
Brief Title: Clinical Course of Cirrhotic Patients With Portal Vein Thrombosis Treated With TIPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, MD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: TIPS-NEOPORTA
Record Dates: First submitted 2017-01-23; First posted 2017-01-26 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Portal Vein Thrombosis
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 3 capillary blood tubes of 4.0 ml Inflammation cytokines will be analyzed (IL-1, IL-6, FNTa)

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt

SUMMARY:
Portal vein thrombosis (PVT) is defined as an obstruction of the portal vein. The prevalence of PVT is 10-25% and incidence is about 16% in cirrhotic patients. PVT leads to increased intrahepatic resistance, decreased portal velocities, splanchnic vasodilatation, and stagnant flow.

Portal vein recanalization (PVR) with transjugular intrahepatic portosystemic shunt (TIPS) is aimed at restoring main portal vein (PV) flow in chronic PVT. In this study, we will review the safety and outcomes of this approach.

DETAILED DESCRIPTION:
Portal vein thrombosis (PVT) is a fairly common complication of liver cirrhosis. Importantly, occlusive PVT might influence the prognosis of patients with cirrhosis. Transjugular intrahepatic portosystemic shunt (TIPS) has been reported to be an effective treatment of PVT in cirrhosis, with the advantage of avoiding the risk of bleeding linked to anticoagulation. In this study, we will evaluate the outcome of TIPS for PVT in patients with and without cirrhosis and determinate survival.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Liver cirrosis or non-cirrhotic patients
* Portal vein thrombosis (degree of vessel obstruction > 50%)

Exclusion Criteria:

* Active variceal bleeding
* Prior history of TIPS placement or shunt surgery
* Concomitant renal insufficiency
* Severe cardiopulmonary diseases
* Uncontrolled sepsis Serious medical conditions which may reduce the life expectancy
* Contraindications for TIPS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with portal vein thrombosis and with or without liver cirrhosis
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Outcome of TIPS for PVT in patients with and without cirrhosis | 5 years
  Clinical evolution after placement of TIPS

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubiran; Aldo Torre Delgadillo, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico